CLINICAL TRIAL: NCT05036083
Title: Added Value of Contrast Enhanced Mammography for Breast Cancer Staging in Patients Referred for a Second Opinion to a Tertiary Cancer Center
Brief Title: Contrast-Enhanced Mammography for Breast Cancer Staging in Patients Referred for a Second Opinion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-1267; NCI-2021-08979 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1267 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Breast Carcinoma; Invasive Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic (CEM, DBT, medical record) (Experimental): Patient receive iodinated contrast agent IV and undergo CEM. Patients who have not undergone DBT as part of their screening or diagnostic imaging within 3 month, undergo DBT. Patients medical records are reviewed.
  Interventions: Procedure: Contrast-Enhanced Mammography; Procedure: Digital Tomosynthesis Mammography; Other: Electronic Health Record Review; Drug: Iodinated Contrast Agent

INTERVENTIONS:
Procedure: Contrast-Enhanced Mammography — Undergo CEM
  Other Names: CEM
Procedure: Digital Tomosynthesis Mammography — Undergo DBT
  Other Names: DBT; Digital Breast Tomosynthesis; Digital Tomosynthesis of the Breast
Other: Electronic Health Record Review — Medical records reviewed
Drug: Iodinated Contrast Agent — Given IV
  Other Names: Iodinated Contrast Dye; Iodine-containing Contrast Media

SUMMARY:
This clinical trial investigates contrast-enhanced mammography (CEM) in detecting breast cancer. CEM is similar to standard mammography, but it includes an injection of an iodine-based contrast, which makes tissue and blood vessels more visible in scans. Diagnostic procedures, such as CEM, may increase the chance of finding breast cancers and decrease the risk of having unnecessary biopsies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the accuracy of CEM and low energy (LE) images (equivalent of full field digital mammogram [FFDM] as the standard of care) for the detection of additional cancer sites in the affected breast and in the contralateral breast.

SECONDARY OBJECTIVES:

I. To evaluate the sensitivity, specificity, positive and negative predictive value of CEM compared to LE CEM images (FFDM equivalent), digital breast tomosynthesis (DBT) and ultrasound for the detection of additional malignant lesions in the ipsilateral and contralateral breast.

II. To evaluate the difference of the index cancer size estimation among CEM, LE images, DBT, and ultrasound compared to pathology measurements as the ground truth.

III. To evaluate the incremental cancer detection rate provided by CEM, DBT, and ultrasound (US) compared to the outside facility (OSF) diagnosis.

EXPLORATORY OBJECTIVES:

I. To evaluate the rate of referral to breast magnetic resonance imaging (MRI) in the study cohort.

II. To evaluate the performance of MRI for breast cancer diagnosis and compare it with other imaging modalities of CEM, LE images, DBT, and US.

III. To evaluate the feasibility of CEM-guided biopsy of CEM-only detected lesions.

OUTLINE:

Patient receive iodinated contrast agent intravenously (IV) and undergo CEM. Patients who have not undergone DBT as part of their screening or diagnostic imaging within 3 month, undergo DBT. Patients medical records are reviewed.

After completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years of age or older with known invasive or in-situ breast cancer (BC) diagnosed at an outside facility and presenting to MD Anderson for staging with imaging
* Female patients 18 years of age or older referred from outside institutions with imaging findings categorized as highly suspicious (Breast Imaging Reporting and Data System [BI-RADS] 5 or 4C) on outside imaging or on rereview by MD Anderson's radiologists and referred for staging at MD Anderson Cancer Center (MDACC)
* Willingness to participate in the study and ability to provide informed consent

Exclusion Criteria:

* Breast surgery within 6 months
* Known allergy to iodine-containing contrast agents
* History of anaphylactic reaction to any substance that required hospitalization or IV placement
* Renal insufficiency; hyperthyroidism
* Detection of non-breast primary or metastatic cancer in the breast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olena Weaver, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible and interested subjects will be consented for study participation. A research staff member who is trained in the informed consent process will explain the study, invite the patients to enroll, and obtain the informed consent of women who wish to participate. Subjects may be enrolled using the approved MD Anderson procedures for remote consenting.
Groups:
- Contrast Enhanced Mammography for Breast Cancer Staging in Patients Referred for Second Opinion: * Female patients with known invasive or in-situ breast cancer diagnosed at an outside facility and presenting to MD Anderson for staging with imaging.
  * Female patients referred from outside institutions with imaging findings categorized as highly suspicious (BI-RADS 5 or 4C) on outside imaging or on re-review by MD Anderson's radiologists, and referred for staging at MDACC.
Period: Overall Study
Arm/Group | Contrast Enhanced Mammography for Breast Cancer Staging in Patients Referred for Second Opinion
Started | 89
Completed | 83
Not Completed | 6
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Labs outside instition parameter, eGFR | 3
Not completed — IV not sustainable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Contrast Enhanced Mammography for Breast Cancer Staging in Patients Referred for Second Opinion
Number analyzed (Participants) | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 72
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 65
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 89

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of CEM for Incremental Cancer Detection in the Ipsilateral and Contralateral Breasts.
Description: Rate of malignancy in lesions de-novo detected on CEM at MDACC and not detected on outside facility imaging. New non-index lesions detected on CEM that had a benign/malignant outcome on image-guided biopsy, surgery, or had a 24-month imaging follow-up with no cancer development (lesion-level evaluation)
  *Index lesion was defined as follows: A) Known cancer detected at an outside facility B) Highly suspicious imaging lesion detected at an outside facility, for which a consultation was requested
Time Frame: One timepoint (at presentation) for lesion characterization with 24 month follow-up for outcome data collection
Measure: Number; unit: % of malignancy in new CEM lesions
Units Other Than Participants: Total number of lesions
Arm/Group | Contrast Enhanced Mammography for Breast Cancer Staging in Patients Referred for Second Opinion
Number analyzed (Participants) | 83
Number analyzed (Total number of lesions) | 164
% of malignancy in new CEM lesions | 41.4

2. Secondary Outcome: Sensitivity, Specificity, Positive and Negative Predictive Value of CEM: RC (Recombined Images) and LE (Low Energy) Images, DBT (Digital Breast Tomosynthesis), and Ultrasound Compared to Pathology as the Ground Truth.
Description: Fraction of malignant lesions detected by each component of CEM
Time Frame: At presentation, Day 1
Measure: Number; unit: lesions
Units Other Than Participants: Total number of lesions
Arm/Group | Contrast Enhanced Mammography for Breast Cancer Staging in Patients Referred for Second Opinion
Number analyzed (Participants) | 83
Number analyzed (Total number of lesions) | 164
lesions
  Total number of detected lesions (index and non-index) | 164
  Malignant index and non-index lesions | 126
  Benign index and non-index lesions | 32
  High-risk lesions | 6
  RC-only detected malignant lesions | 20
  LE+RC detected malignant lesions | 103
  LE-only detected malignanct lesions | 3

3. Secondary Outcome: Percentage of Lesions That Appeared Larger on CEM
Description: Largest measurements in imaging were compared to the largest measurements in pathology and the size difference of 5mm or more was considered significant. Fraction of patients in whom CEM detected an increase in lesion size of 5 mm or more was reported and analyzed.
Time Frame: One timepoint- at presentation
Measure: Number; unit: % of malignant lesions larger on CEM
Units Other Than Participants: Total number of lesions
Arm/Group | Contrast Enhanced Mammography for Breast Cancer Staging in Patients Referred for Second Opinion
Number analyzed (Participants) | 83
Number analyzed (Total number of lesions) | 164
% of malignant lesions larger on CEM | 28

4. Secondary Outcome: Incremental Cancer Detection Rate Provided by CEM, DBT and US Compared to Outside Imaging
Description: Percentage of patients with a change in the number of cancers sites (unifocal, multifocal, or bilateral) compared to outside facility imaging interpretation
Time Frame: 1 timepoint at presentation
Population: Patients who had additional malignant lesions detected as a result of CEM work-up
Measure: Count of Participants; unit: Participants
Arm/Group | Contrast Enhanced Mammography for Breast Cancer Staging in Patients Referred for Second Opinion
Number analyzed (Participants) | 83
Participants
  Patients with unifocal cancer as detected at outside imaging | 68
  Patients with unifocal cancer after MDACC work-up | 50
  Patients with unknown staging as presented at outside imaging | 3
  Patients with unknown staging after MDACC work-up | 0
  Mutlicentric/miultifocal cancer as detected at outside imaging | 11
  Mutlicentric/miultifocal cancer after MDACC work-up | 27
  Patients with bilateral cancer at outside imaging | 1
  Patients with bilateral cancer after MDACC work-up | 6

5. Secondary Outcome: Rate of Malignancy
Description: Rate of RC-only detected malignancy, LE+RC detected malignancy, LE-only detected malignancy
Time Frame: One timepoint (at presentation) for lesion characterisation with 24 mo follow-up for outcome data collection
Measure: Number; unit: percentage of malignancy
Units Other Than Participants: Total number of lesions
Arm/Group | Contrast Enhanced Mammography for Breast Cancer Staging in Patients Referred for Second Opinion
Number analyzed (Participants) | 83
Number analyzed (Total number of lesions) | 164
percentage of malignancy
  Rate of RC-only detected malignancy (%) | 16
  Rate of LE+RC detected malignancy (%) | 82
  Rate of LE-only detected malignancy (%) | 8

6. Other Pre Specified Outcome: Rate of Breast MRI Utilization and the Corresponding Diagnosis in the Study Cohort.
Description: Percentage of patients who underwent both CEM and MRI
Time Frame: One timepoint for CEM data (at presentation) +/- 2 month (4 month total) for MRI
Population: Study patients who underwent both breast MRI and CEM. The fraction of the patients with MRI prompting a change in management
Measure: Count of Participants; unit: Participants
Arm/Group | Contrast Enhanced Mammography for Breast Cancer Staging in Patients Referred for Second Opinion
Number analyzed (Participants) | 83
Participants
  Patients with breast MRI | 33
  MRI changed management | 20

7. Other Pre Specified Outcome: The Fraction of CEM Biopsies That Achieve Adequate Sampling of the Target.
Description: Patients who required a CEM-guided biopsy and successfully underwent it with adequate tissue sampling. Percentage of all non-index CEM lesions that required a CEM biopsy.
Time Frame: Two timepoints- at first CEM imaging presentation and at CEM-guided biopsy (within 2 months)
Measure: Number; unit: percentage of successful CEM biopsies
Units Other Than Participants: Lesions
Arm/Group | Contrast Enhanced Mammography for Breast Cancer Staging in Patients Referred for Second Opinion
Number analyzed (Participants) | 83
Number analyzed (Lesions) | 53
percentage of successful CEM biopsies
  Fraction of non-index lesions recommended for a CEM-guided biopsy (%) | 15
  Fraction of successful CEM-guided biopsies (%) | 100

ADVERSE EVENTS:
Time Frame: At presentation, Day 1
Arm/Group | Contrast Enhanced Mammography for Breast Cancer Staging in Patients Referred for Second Opinion
All-Cause Mortality (participants affected / at risk) | 0/89
Serious Adverse Events (participants affected / at risk) | 0/89
Other Adverse Events (participants affected / at risk) | 2/89
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Contrast Enhanced Mammography for Breast Cancer Staging in Patients Referred for Second Opinion (N=89)
Saline flush extravasation (General disorders) | 1
Mild nausea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT05036083/Prot_SAP_000.pdf